CLINICAL TRIAL: NCT05203705
Title: Efficacy and Safety of SHR2285 Tablets Following Multiple Oral Administrations in Patients Undergoing Elective Total Knee Arthroplasty: a Multicenter, Randomized, Positive-controlled Phase II Clinical Study
Brief Title: Clinical Study on the Efficacy and Safety of Multiple Oral Administrations of SHR2285 Tablets in Patients Undergoing Elective Total Knee Arthroplasty
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Adjustment of the sponsor's R&D strategy
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR2285-201
Record Dates: First submitted 2022-01-20; First posted 2022-01-24 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Prevention of Venous Thrombosis After TKA
MeSH Terms: interventions — Enoxaparin

STUDY DESIGN:
Intervention Model Description: SHR2285 tablets compared with Enoxaparin
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Treatment group 1 (Experimental): SHR2285 tablet; dose 1
  Interventions: Drug: SHR2285 tablet
- Treatment group 2 (Experimental): SHR2285 tablet; dose 2
  Interventions: Drug: SHR2285 tablet
- Treatment group 3 (Experimental): SHR2285 tablet; dose 3
  Interventions: Drug: SHR2285 tablet
- Treatment group 4 (Experimental): SHR2285 tablet; dose 4
  Interventions: Drug: SHR2285 tablet
- Treatment group 5 (Active Comparator): Enoxaparin
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: SHR2285 tablet — SHR2285 tablet; dose 1, for 12 days
  Arms: Treatment group 1
Drug: SHR2285 tablet — SHR2285 tablet; dose 2, for 12 days
  Arms: Treatment group 2
Drug: SHR2285 tablet — SHR2285 tablet; dose 3, for 12 days
  Arms: Treatment group 3
Drug: SHR2285 tablet — SHR2285 tablet; dose 4, for 12 days
  Arms: Treatment group 4
Drug: Enoxaparin — Enoxaparin, for 12 days
  Arms: Treatment group 5

SUMMARY:
This study is a multi-center, randomized, open-label, double-blind, positive-controlled phase II clinical study evaluating the efficacy and safety of different doses of SHR2285 tablets vs. enoxaparin for the prevention of postoperative venous thromboembolism in patients undergoing elective unilateral total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the study procedures and methods, voluntarily participate in the study, and sign the written informed consent form (ICF);
2. Scheduled to undergo elective unilateral total knee arthroplasty;
3. Males or females aged 40-75 years.

Exclusion Criteria:

1. Weighing less than 40 kg or greater than 135 kg;
2. Allergic to contrast agents rendering the patient unable to undergo venous angiography of the lower extremities; allergic to enoxaparin or any of the ingredients listed in the package insert thereof; allergic to the investigational product or any of the ingredients thereof;
3. With malignant tumors that still require medical intervention; except for radically treated non-melanoma skin cancer, basal cell carcinoma or squamous cell skin cancer, or cervical carcinoma in situ;
4. With a history of major liver disease within 1 year;
5. With myocardial infarction, transient ischemic attack, or ischemic stroke within 6 months.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
Number of patients with confirmed composite endpoint | Day 12
  Occurrence of confirmed composite endpoint of asymptomatic deep vein thrombosis (DVT), confirmed symptomatic/non-symptomatic venous thromboembolic events (VTE), non-fatal pulmonary embolism (PE) or all-cause deaths
Number of patients with composite bleeding | Day 12
  Occurrence of confirmed composite endpoint of major bleeding and clinically relevant non-major (CRNM) bleeding events

SECONDARY OUTCOMES:
Number of patients with composite venous thromboembolic events (VTE) | Day 1 to Day 12
  Occurrence of confirmed composite endpoint of asymptomatic deep vein thrombosis (DVT), Confirmed symptomatic/non-symptomatic venous thromboembolic events (VTE), non-fatal pulmonary embolism (PE) ,all-cause deaths
Number of patients with composite venous thromboembolic events (VTE) | Day 1 to Day 42
  Occurrence of confirmed composite endpoint of asymptomatic deep vein thrombosis (DVT), Confirmed symptomatic/non-symptomatic venous thromboembolic events (VTE), non-fatal pulmonary embolism (PE) ,all-cause deaths

CONTACTS AND LOCATIONS:
Locations (1):
- Perking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided